CLINICAL TRIAL: NCT06659042
Title: A Prospective, Single-arm Phase II Study of the Efficacy and Safety of Tislelizumab in Combination With Chemotherapy Perioperative Treatment for Resectable II-IIIB(N2) KRAS-mutated Nonsquamous Non-small Cell Lung Cancer
Brief Title: Perioperative Tislelizumab for Resectable II-IIIB(N2) KRAS-mutated Nonsquamous Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Feng Yao, Vice President of Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024IIT-145
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer, Non-Small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab plus platinum doublet chemotherapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed Disodium

INTERVENTIONS:
Drug: Tislelizumab — administered via Intravenous (IV) injection
Drug: Cisplatin — administered via IV infusion
Drug: Carboplatin — administered via IV infusion
Drug: Pemetrexed Disodium — administered via IV infusion

SUMMARY:
The primary objective of the perioperative study is to evaluate pathological complete response in resectable II-IIIB(N2) KRAS-mutated nonsquamous non-small cell lung cancer participants receiving tislelizumab plus platinum-based doublet chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent (ICF) and able to understand and comply with the study requirements and assessment schedule.
2. Male or female aged ≥18 years at the time of signing the ICF.
3. Histologically or cytologically confirmed stage II-IIIB (N2) non-squamous non-small cell lung cancer (NSCLC) (AJCC 8th edition).
4. With Known KRAS gene mutation.
5. Evaluated by medical and surgical discussion to be eligible for R0 resection with curative intent prior to study enrollment.
6. At least one measurable lesion as defined by RECIST v1.1.
7. Eligible to receive platinum-based doublet chemotherapy.
8. ECOG performance status score ≤ 1.
9. Adequate organ function during the screening period
10. Good cardiopulmonary function, meeting the requirements for surgical resection with curative intent.
11. Patients of childbearing potential must be willing to use effective contraception during the study and for 120 days after the last dose of tislelizumab.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for enrollment:

1. Previously received any treatment for the current lung cancer, including radiotherapy and all systemic anti-tumor treatments, including chemotherapy, immunotherapy, targeted therapy, or anti-angiogenic therapy.
2. Presence of locally advanced, unresectable disease, regardless of disease stage or presence of metastases.
3. Received other approved systemic immunomodulatory agents (including but not limited to interferon, interleukin-2, tumor necrosis factor, thymosin α1, and thymalfasin) within 4 weeks prior to the first dose.
4. Used any herbal medicine to control cancer within 14 days prior to the first dose of the study drug.
5. Received live or attenuated live vaccines within 4 weeks prior to enrollment or expected to require live or attenuated live vaccines during the study or within 5 months after the last dose of tislelizumab.
6. Any condition requiring systemic corticosteroid therapy (prednisone or equivalent >10 mg/day) or other immunosuppressive therapy within 14 days prior to the first dose of the study drug, which the investigator believes may affect the study treatment.
7. Active autoimmune disease requiring systemic treatment, which the investigator believes may affect the study treatment.
8. Interstitial lung disease, non-infectious pneumonitis, or uncontrolled other diseases, including diabetes, pulmonary fibrosis, acute lung disease, etc., which the investigator believes may affect the study treatment.
9. History of major diseases or clinical manifestations that may affect organ system function, which the investigator believes may affect the study treatment.
10. Severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral treatment within 14 days prior to the first dose of the study drug (including tuberculosis infection, etc.).
11. Known history of human immunodeficiency virus (HIV) infection.
12. Previously undergone allogeneic stem cell transplantation or organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Up to 3 months following completion of neoadjuvant treatment

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | Up to 3 months following completion of neoadjuvant treatment
Objective Response Rate (ORR) | Up to 3 years
Event-free survival (EFS) | Up to 3 years
Overall survival (OS) | Up to 3 years
Number of participants experiencing treatment-emergent adverse events (TEAEs) | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No